CLINICAL TRIAL: NCT06106516
Title: Vital Sign Monitor Device Validation - WARD
Acronym: ViVa-WARD
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Professor, Rigshospitalet, Denmark
Other Study IDs: WZ-23050470
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Surgery-Complications; Medical Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: novel vital sign monitor — Devices that are to be introduced into the clinic but where data from clinical relevant conditions such as complications are lacking to assess the validity under clinical conditions

SUMMARY:
Aim: to assess the validity of CE/FDA approved vital sign monitor devices for clinical use in clinical setting.

Patients: up to 1000 medical and/or surgical patients will be included Intervention: Studies with various wirless or novel vital sign monitor devices control: Golden standard measurements or clinical standard devices Outcome: Agreement assessed by bias and limits of agreement between Intervention and control device.

DETAILED DESCRIPTION:
Aim: to assess the validity of CE/FDA approved vital sign monitor devices for clinical use in clinical setting.

Patients: up to 1000 medical and/or surgical patients will be included. Intervention: Studies with various wireless or novel vital sign monitor devices control: Golden standard measurements or clinical standard devices Outcome: Agreement assessed by bias and limits of agreement between Intervention and control device. Other statistical assessments of agreement may be chosen as secondary outcomes, dependent on the data-structure

Setting: the study will be carried out in up to 76 hours with collection of vital sign data pre-, intra or postoperatively.

ELIGIBILITY:
No inclusion or exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Humans with or without medical or surgical complications in or out of hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between vital sign data from novel device and golden standard | 76 hours
  agreement between novel device and golden standard or clinical standard devices, assess by bias and limits of agreement

SECONDARY OUTCOMES:
Description of data from novel device and golden standard | 76 hours
  descriptive statistics using parametric or non-parametric statistics where appropriate

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Eske Kvanner Aasvang, Copenhagen
  - Bispebjerg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided
data can be shared upon reasonable request